CLINICAL TRIAL: NCT04338139
Title: Influence of Bio-Oss Collagen Grafting at Implant Placement on Buccal Bone Volume Regeneration: a Human Study
Brief Title: Influence of Bio-Oss Collagen Grafting at Implant Placement on Buccal Bone Volume Regeneration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USJ-2019-112
Record Dates: First submitted 2020-04-05; First posted 2020-04-08 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Bone Regeneration
MeSH Terms: interventions — Bone Regeneration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bio-oss Collagen (Experimental): 90% xengeneic bovine bone partciles + 10% collagen type I
  Interventions: Procedure: bone regeneration

INTERVENTIONS:
Procedure: bone regeneration — bone regeneration using bio-oss collagen

SUMMARY:
to validate the capacity of bio-oss collagen (xenograft block+ collagen type I) placed solely without a membrane on a thin (0.5-1.8mm) buccal bone wall after delayed implant placement to regenerate bone volume. 30 patients requiring dental implants and presenting a deficient bone ridge (a ridge with reduced marginal bone width ≤ 2mm) were selected. The bone regeneration technique used in this study:

* Pre-operatively:

  * cone beam computed tomography CBCT
  * 1 minute mouthwash with a 0.12% Chlorhexidine solution
  * Full thickness muco-periosteal flap and ridge curettage.
  * Drilling and implant placement (any implant system)
  * Adjustment and placement of the "Bio-Oss Collagen" in the regeneration site without a fixation membrane.
  * Hermetic wound closure with U-shaped and simple stitches using 5/0 and 6/0 PGA resorbable material.
* Post-operatively:

  * Medication:

    * Amoxicilline (1g) or Clindamycine (300mg)
    * Analgesic, (paracetamol + codeine)
  * Mouthwash with a solution of 0.12% Chlorhexidine
  * cone beam computed tomography CBCT

    * 4 months postoperatively: CBCT

Bio-oss collagen is placed on the buccal side after implant placement and adapted to have the bone defect morphology. the full thickness flap is then closed without membrane placement and the bone bock is fixed in place through sutures only. CBCT images were taken immediately postoperatively and at 4 months after bone grafting. Imaging superposition (on ITK software) and measurements of buccal bone gain were effectuated to evaluate the efficiency of this regeneration technique. evaluation of buccal bone regeneration through linear radiographic measurements and evaluation of the % of grafted bone resorption will indicate the success of this technique

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Smoking <10 cigarettes/day (Light smoker)
* Good general health.
* Absence of acute infection: edema, suppuration, abscess, spontaneous bleeding.

Exclusion Criteria:

* A pregnant or nursing mother
* Pathologies that may impair bone healing: diabetes, autoimmune diseases, corticosteroids, chemotherapy.

Orthodontic treatment in progress or planned

- Adjacent risk teeth

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
linear measurements on the superimposed CBCTs of the buccal bone width gain at different locations | 1 year
  cbct radiographic measurements

SECONDARY OUTCOMES:
linear measurements of the amount of grafted bone resorption | 1 year
  cbct radiographic measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Saint-Joseph University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
article publication
Time Frame: 1 year
Access Criteria: article publication